CLINICAL TRIAL: NCT06551155
Title: Identification, Monitoring, and Classification of Patients at Risk of Osteoporosis and Fractures Using a Method Based on the Use of Mononuclear Cells From Peripheral Blood
Brief Title: Peripheral Mononuclear Cells to Screen, Monitor and Stratify the Population at Risk of Osteoporosis and Fractures
Acronym: DISCERN
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: Azienda Ospedaliero Universitaria Policlinico G.Rodolico - San Marco (Unknown)
Responsible Party: Sponsor
Other Study IDs: DISCERN
Record Dates: First submitted 2024-08-09; First posted 2024-08-13 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Osteoporosis; Osteopenia; Osteoporosis Fracture
Keywords: peripheral blood mononuclear cells; screening; diagnosis
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic; Osteoporotic Fractures; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Healthy patients: Patients with available DXA results, at risk and in periodic follow-up and/or attending outpatient visits for preventive screening
  Interventions: Diagnostic Test: Vitality and biological activity of peripheral blood mononuclear cells (PBMCs)
- Osteopenic patients: Patients with available DXA results, enrolled during outpatient visits and/or emergency room and/or hospital admissions
  Interventions: Diagnostic Test: Vitality and biological activity of peripheral blood mononuclear cells (PBMCs)
- Non-fractured osteoporotic patients: Patients with available DXA results, enrolled during outpatient visits and/or emergency room and/or hospital admissions
  Interventions: Diagnostic Test: Vitality and biological activity of peripheral blood mononuclear cells (PBMCs)
- Fractured osteoporotic patients: Patients with available DXA results or prescribed as per clinical practice, enrolled during hospital admissions
  Interventions: Diagnostic Test: Vitality and biological activity of peripheral blood mononuclear cells (PBMCs)

INTERVENTIONS:
Diagnostic Test: Vitality and biological activity of peripheral blood mononuclear cells (PBMCs) — Diagnostic test based on the vitality and biological activity of peripheral blood mononuclear cells (PBMCs) tested analyzing approximately 2-5 mL of blood from healthy patients and from osteopenic and osteoporotic (both fractured and non-fractured) patients of both genders

SUMMARY:
Osteoporosis (OP) is one of most common age-associated and chronic metabolic bone diseases, featured by a decrease of bone mineral density (BMD) that increases the risk of bone fractures.OP guidelines agree that Dual-X-ray Absorptiometry (DXA) is the gold standard for BMD assessment, but for the different OP stages screening and diagnosis, BMD by itself is not an accurate predictor. Thus, OP is often misdiagnosed. Aim of the this study is to improve a tool for OP diagnosis based on the ability of circulating peripheral blood mononuclear cells (PBMCs) to maintain or not their in vitro viability (IRCCS Istituto Ortopedico Rizzoli European patent n.3008470 March 21, 2018) for the measurement of the different OP severity levels, also considering specific gender related differences.

DETAILED DESCRIPTION:
Inadequate assessment, diagnosis, and stratification of patients with bone mass loss can lead to an increased risk of osteoporotic fractures. Therefore, alternative and advanced methods to support screening and diagnosis of osteoporosis (OP) are becoming increasingly essential, particularly considering specific gender differences. In this context, evaluating new methods and innovative techniques is a global challenge. To address this challenge, in 2018, the IRCCS Istituto Ortopedico Rizzoli (IOR) filed a European patent (European Patent No. 3008470, March 21, 2018; Inventors: Fini M, Giardino R, Salamanna F) related to an in vitro method for correlating the vitality of peripheral blood mononuclear cells (PBMCs) with bone metabolism alterations and OP through simple optical microscope observation. Additionally, specific gender-related differences have been observed in the number, size, differentiation time, and gene and protein expression profiles of PBMCs from osteoporotic patients of different sexes. In this context, the purpose of this study is to fully expand and develop the patent filed by IRCCS IOR in 2018 in order to: a) improve the understanding of the mechanisms of action and observed behavior in PBMCs on which the IOR patent is based; b) correlate the in vitro behavior of PBMCs with different levels of bone metabolism alteration (from osteopenia to fragility fractures); c) evaluate the correlation between the Dual-X-ray Absorptiometry (DXA) T-score and other blood factors related to OP (parameters related to platelets, pro- and anti-inflammatory cytokines, lymphocyte subpopulations) with the in vitro behavior of PBMCs in the presence of different levels of bone metabolism alteration, considering specific gender differences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients (at risk and undergoing periodic follow-up and/or attending outpatient visits for preventive screening)
* Osteopenic patients with an available DXA
* Osteoporotic patients (fractured and non-fractured) with an available DXA or, for fractured patients, a DXA prescribed as part of clinical practice
* Aged ≥ 40 years of both sexes
* Body Mass Index (BMI) between 18.5 and 29.9

Exclusion Criteria:

* Hematopoietic system disorders (hemolytic, aplastic, and neoplastic anemias)
* Coagulation disorders (hereditary or secondary to other disorders)
* Infections (including HIV-HBV-HCV positivity)
* Neoplastic diseases (primary and/or secondary tumors)
* Pregnancy or breastfeeding
* Alcohol consumption (>20 g of alcohol per day currently or in the past)
* Smoking (>10 cigarettes per day, currently or in the past)
* Diabetes
* Treatment with therapeutic agents that may interfere with hematopoiesis (corticosteroids, immunosuppressive agents, cytotoxic drugs)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy patients (at risk and undergoing periodic follow-up and/or attending outpatient visits for preventive screening), osteopenic patients, and those with osteoporosis (fractured and non-fractured) with an available DXA or, for fractured patients, a DXA prescribed as part of clinical practice, aged ≥ 40 years of both sexes, with a Body Mass Index (BMI) between 18.5 and 29.9.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-08-05 (Actual); Primary Completion 2026-01-05 (Estimated); Study Completion 2026-08-05 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity | January 2026
  The primary outcome is to determine the sensitivity and specificity of the in vitro behavior (vitality, number, size, and differentiation) of PBMCs (peripheral blood mononuclear cells) in relation to different levels of bone metabolism alteration (ranging from osteopenia to fragility fractures).

SECONDARY OUTCOMES:
Correlation | January 2026
  The secondary outcomes include the evaluation and correlation of BMD via DXA T-score, vitality, number, size, and differentiation of PBMCs, T lymphocyte subpopulations, pro- and anti-inflammatory factors, platelet-related parameters, and the expression of biochemical markers of bone turnover in blood and serum samples from healthy individuals, as well as from osteopenic and osteoporotic patients (both fractured and non-fractured).

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Ortopedico Rizzoli, Bologna
  - Azienda Ospedaliero Universitaria Policlinico G.Rodolico - San Marco, Catania

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Salamanna F, Maglio M, Giavaresi G, Pagani S, Giardino R, Fini M. In vitro method for the screening and monitoring of estrogen-deficiency osteoporosis by targeting peripheral circulating monocytes. Age (Dordr). 2015 Aug;37(4):9819. doi: 10.1007/s11357-015-9819-4. Epub 2015 Aug 7. PMID 26250906
- [Result] Salamanna F, Maglio M, Borsari V, Giavaresi G, Aldini NN, Fini M. Peripheral Blood Mononuclear Cells Spontaneous Osteoclastogenesis: Mechanisms Driving the Process and Clinical Relevance in Skeletal Disease. J Cell Physiol. 2016 Mar;231(3):521-30. doi: 10.1002/jcp.25134. Epub 2015 Sep 9. PMID 26284737
- [Result] Salamanna F, Giardino R, Fini M. Spontaneous osteoclastogenesis: Hypothesis for gender-unrelated osteoporosis screening and diagnosis. Med Hypotheses. 2017 Nov;109:70-72. doi: 10.1016/j.mehy.2017.09.028. Epub 2017 Sep 28. PMID 29150298
- [Result] Salamanna F, Maglio M, Sartori M, Tschon M, Fini M. Platelet Features and Derivatives in Osteoporosis: A Rational and Systematic Review on the Best Evidence. Int J Mol Sci. 2020 Mar 4;21(5):1762. doi: 10.3390/ijms21051762. PMID 32143494
- [Derived] Salamanna F, Brogini S, Di Martino A, Baldini N, Gaudio A, Castellino P, Contartese D, Di Censo C, Giavaresi G, Faldini C, Fini M. Sustainable innovation with a method based on peripheral mononuclear cells to screen, monitor and stratify the population at risk of osteoporosis and fractures - a multicenter cross-sectional trial protocol. Front Endocrinol (Lausanne). 2025 Oct 2;16:1647800. doi: 10.3389/fendo.2025.1647800. eCollection 2025. PMID 41113706